CLINICAL TRIAL: NCT00106652
Title: Environmental Factors in the Etiology of Autism
Brief Title: Childhood Autism Risks From Genetics and the Environment (The CHARGE Study)
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Collaborators: University of California, Davis (Other); University of California, Los Angeles (Other)
Other Study IDs: 11269-CP-001; 200210574-4
Record Dates: First submitted 2005-03-28; First posted 2005-03-29 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Autism; Developmental Disabilities
Keywords: autism; neurodevelopment; neurotoxicology; perinatology; teratology
MeSH Terms: conditions — Autistic Disorder; Developmental Disabilities

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
The purpose of this study is to understand how genes, environment, and the interplay between the two, influences the development of autism and other neurodevelopmental disorders.

DETAILED DESCRIPTION:
The causes and contributing factors for autism are poorly understood. Evidence suggests that incidence is increasing, but diagnostic changes and improvements may be playing a role. Both genetic and environmental factors appear to play a role. Autopsy studies demonstrate structural changes in the brain and clinical investigations reveal neurophysiologic differences in information processing in autistic versus normal children. Members of our team recently demonstrated altered levels of certain neuropeptides at birth in children who later developed autism.

This case-control study is the first large-scale epidemiologic investigation of underlying causes for autism and triggers of regression. This study capitalizes on the strengths of the case-control design, which is well suited to examine a broad array of factors for rare conditions that are thought to be multifactorial. Comparisons will be made with both general population controls and mentally retarded children.

The aims are to assess the influence of exogenous exposures, the role of susceptibility factors, and the interplay between these two in the etiology of autism and its phenotypic variation. Chemicals with known or suspected neurodevelopmental toxicity, such as PCB's, certain pesticides, and metals, are being investigated. This study pursues several hypotheses that have recently gained attention, including the combined measles, mumps, rubella vaccine and mercury present in vaccines given during infancy and early childhood. Additionally, biochemical susceptibility is examined through characterization of metabolic, immunologic, and neuronal gene expression profiles and genetic polymorphisms.

ELIGIBILITY:
Inclusion Criteria:

* Children between 2 and 5 years old
* Born in California
* Parents must speak either English or Spanish
* Children must be living with at least one biologic parent

Exclusion Criteria:

* Children not meeting eligibility criteria listed above
* Children not residing in selected geographical areas (please contact for more information about specific study locations)

Ages: 24 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2000 (Estimated)
Dates: Start 2001-09; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isaac N. Pessah, Ph.D., Principal Investigator — University of California, Davis; Irva Hertz-Picciotto, Ph.D., Study Director — University of California, Davis
Locations (1):
- University of California, Davis, California, United States

REFERENCES:
- See also: click for more information about this study: Childhood Autism Risks from Genetics and the Environment — http://beincharge.ucdavis.edu
- See also: click here for more information about the UC Davis M.I.N.D. Institute — http://www.ucdmc.ucdavis.edu/mindinstitute